CLINICAL TRIAL: NCT01305070
Title: Femoral Artery In-Stent Restenosis (FAIR) Trial
Brief Title: Standard Balloon Angioplasty Versus Angioplasty With a Paclitaxel-eluting Balloon for Femoral Artery In-stent Restenosis
Acronym: FAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical Care Center Prof. Mathey, Prof. Schofer, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAIR 3.0
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2013-04

CONDITIONS: Peripheral Vascular Disease
Keywords: Standard balloon angioplasty; POBA; Angioplasty with paclitaxel-eluting balloon; Superficial femoral artery
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standart balloon angioplasty (Active Comparator): Admiral Xtreme, Invatec
  Interventions: Device: Admiral Xtreme
- Paclitaxel-eluting balloon arm (Active Comparator): In.Pact Admiral, Invatec
  Interventions: Device: In.Pact Admiral

INTERVENTIONS:
Device: Admiral Xtreme — For balloon angioplasty of in-stent restenosis in the superficial femoral artery
  Other Names: Admiral Xtreme, Invatec
  Arms: Standart balloon angioplasty
Device: In.Pact Admiral — For balloon angioplasty of in-stent restenosis in the superficial femoral artery
  Other Names: In.Pact Admiral, Invatec
  Arms: Paclitaxel-eluting balloon arm

SUMMARY:
Comparison of recurrent-restenosis rates 6 months after angioplasty of in-stent restenoses or in-stent reocclusions in the superficial femoral artery (SFA) using either a standard balloon (Admiral Xtreme, Invatec) or a paclitaxel-eluting balloon (In.Pact™ Admiral, Invatec).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 years old.
2. Patient must sign informed consent form.
3. Patient must agree to participate in the study and comply with follow-up requirements.
4. Clinically, all patients must be in Rutherford category 2 to 4.

   Angiographic Inclusion Criteria:
5. Planned angioplasty of in-stent restenoses (degree of stenosis 70-100%) within the SFA. The target lesion must not extend beyond the stent margins. In cases of two or more stenotic regions within the stented segment, these are considered separate lesions if there is a nonstenotic or only mildly stenotic (< 30%) segment of at least 2 cm in length between them. Otherwise, they are considered a single lesion. In case of separate lesions, only the proximal lesion will be taken as the target lesion!
6. The length of the in-stent lesion should be at least 1 cm and maximally 20 cm (measurement by radiopaque ruler).
7. The degree of target lesion stenosis must be determined by pre-interventional duplex ultrasound.
8. The target lesion region starts at the origin of the SFA and ends distally at the femoropopliteal crossover (crossing by SFA of medial rim of femur in the PA projection).
9. Patency (< 50% stenosis) of popliteal artery and at least 1 infragenicular artery.

Exclusion Criteria:

General:

1. Patient is currently participating in another clinical trial.
2. Pregnancy or pregnancy planned during study duration.
3. Life expectancy less than 1 year.
4. Co-morbidities preventing study participation.
5. Severe coagulation disorders.
6. Current treatment with anticoagulants other than aspirin, ticlopidine, clopidogrel or prasugrel.
7. Active gastric ulcer or gastrointestinal bleeding.
8. Thrombotic occlusion of the target vessel within previous 4 weeks.
9. Treatment of target lesion with laser or atherectomy devices.
10. Dialysis dependency.
11. Manifest hyperthyreosis.
12. Known allergy against contrast agent that cannot be adequately controlled by usual premedication.
13. Known heparin intolerance.
14. Known paclitaxel intolerance.

    Angiographic:
15. Target lesion extends into the popliteal artery.
16. Symptomatic untreated inflow lesion > 50% in ipsilateral iliac arteries. Pretreatment of iliac stenoses is possible.
17. SFA lesions > 50% stenosis proximal and/or distal to the target lesion that require treatment.
18. Target lesion extends beyond the stent margins.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Duplex-ultrasound determined recurrent restenosis in the superficial femoral artery (SFA) | 6 month
  Binary restenosis rate by Duplex-ultrasound >= 50% measured as proximal peak velocity ratio PVR[prox] >= 2.4

SECONDARY OUTCOMES:
Recurrent restenosis within the stent at 12 month | 12 month
  Recurrent restenosis >= 50% measured as proximal peak velocity ratio PVR[prox] >= 2.4
Clinically driven target lesion revascularization (TLR) at 6 and 12 month | 6 and 12 month
Recurrent stenosis >= 70% within the stent at 6 and 12 month | 6 and 12 month
  Recurrent restenosis >= 70% measured as proximal peak velocity ratio PVR[prox] >= 3.4
Clinical and hemodynamic parameters | at 1, 6 and 12 month
  Walking distance, ABI, Rutherford category
Primary angiographic success rate | 12 month
  Angiographic sucess: <50% residual stenosis
Major adverse vascular events (MAVE) | 12 month
Death | 12 month
Impact of "bail-out" stent-in-stent placement on 6-and 12-month end points | 6 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Hans Krankenberg, MD, Principal Investigator — Medical Care Center Prof. Mathey, Prof. Schof Ltd.; Thilo Tübler, MD, Study Chair — Medical Care Center Prof. Mathey, Prof. Schofer
Locations (1):
- Medical Care Center Prof. Mathey, Prof. Schofer, Hamburg, Hamburg, Germany

REFERENCES:
- [Derived] Krankenberg H, Tubler T, Ingwersen M, Schluter M, Scheinert D, Blessing E, Sixt S, Kieback A, Beschorner U, Zeller T. Drug-Coated Balloon Versus Standard Balloon for Superficial Femoral Artery In-Stent Restenosis: The Randomized Femoral Artery In-Stent Restenosis (FAIR) Trial. Circulation. 2015 Dec 8;132(23):2230-6. doi: 10.1161/CIRCULATIONAHA.115.017364. Epub 2015 Oct 7. PMID 26446728